CLINICAL TRIAL: NCT05781880
Title: Efficiency and Safety Evaluation of Normobaric Hyperoxia Stabilizing the Penumbra in Patients With Acute Ischemic Stroke
Brief Title: Normobaric Hyperoxia Stabilizing Ischemic Penumbra
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ji Xunming,MD,PhD (Other)
Responsible Party: Sponsor-Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Organization: Capital Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NBOTIP
Record Dates: First submitted 2023-03-06; First posted 2023-03-23 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Acute Ischemic Stroke
Keywords: Normobaric Hyperoxia; Acute ischemic stroke; penumbra
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes indexes will be assessed by trained neurologists or neuroradiologists who are blinded to the research content or patient grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO group (Experimental): Normobaric hyperoxia (NBO) oxygen group will be given 100% oxgen (10L/min for 4h) via a face mask.
  Interventions: Other: Oxygen 100%
- Control group (Placebo Comparator): Control group will be given nasal oxygen (2L/min for 4h）. All other therapy measures are the same as experimental group.
  Interventions: Other: Oxygen 100%

INTERVENTIONS:
Other: Oxygen 100% — NBO therapy were given 100% oxygen via a face mask (10L/min for 4h)
  Other Names: Normobaric hyperoxia

SUMMARY:
To investigate the safety and efficacy of normobaric hyperoxia (NBO) stabilizing penumbra in acute ischemic stroke patients.

DETAILED DESCRIPTION:
All the enrolled patients were randomly assigned to NBO and control group. NBO group will be given 100% oxygen ( (10L/min for 4h) via a storage oxygen face mask and control group will be given oxygen using nasal oxygen(2L/min for 4h) .

ELIGIBILITY:
Inclusion criteria:

* Age≥18岁
* The signs and symptoms are consistent with anterior circulation infarction, and baseline NIHSS score：6-20
* Level of consciousness on admission：0-1
* mRS score before stroke: 0-1
* Patients who did not receive revascularization therapy
* The time from onset (finally normal) to randomization is less than 24h
* Patients who signed informed consent
* CTA or MRA confirmed internal carotid artery occlusion or M1/M2 segment occlusion of middle cerebral artery
* The low-perfusion area with Tmax>6s was larger than the core infarction, and the mismatch ratio was greater than or equal to 1.8.

Exclusion Criteria:

* Evidence of rapid improvement in neurological function and NIHSS score <6, or spontaneous recanalization before randomization
* The disease affecting assessment of baseline NIHSS score (dementia, epilepsy, neuromuscular disease, or psychiatric disease)
* Symptoms suggesting subarachnoid hemorrhage (even if CT scan is normal)
* Combined with the history, cerebral embolism due to sepsis or infective endocarditis was suspected
* Active or chronic obstructive pulmonary disease, pulmonary fibrosis, pneumonia, pleural effusion, acute respiratory distress syndrome, irregular breathing
* It is necessary to inhale (>3L/min) oxygen to maintain peripheral arterial oxygen saturation (SaO2>95%)
* Anemia or polycythemia vera or other conditions needing emergency oxygen patients
* Patients with upper gastrointestinal bleeding or nausea and vomiting can not complete inhalation oxygen using face mask
* Baseline blood glucose <2.78mmol/L or >22.2mmol/L
* Baseline platelet count <50×109/L
* Hereditary or acquired bleeding tendency, lack of coagulation factor, recent oral anticoagulant INR>3 or PPT more than 3 times
* Unstable vital signs (heart rate ≤50 beats/min or ≥120 beats/min, oxygen saturation ≤90%, R≥30 beats/min or ≤10 beats/min)
* Hypertension not controlled by medication: systolic blood pressure ≥185mmHg, or diastolic blood pressure ≥110mmHg
* Acute myocardial infarction suspected
* Pregnancy,
* Life expectancy <90 days
* Heart, liver and kidney failure
* Magnetic resonance contraindications
* Claustrophobia
* Allergic to contrast media
* Participating in other drug or device research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
changing of penumbra volume from baseline | Day 0
  the comparison of ratio of 4h following randomizing and baseline for penumbra volume between NBO and control group

SECONDARY OUTCOMES:
penumbra volume at 4h following randomizing | Day 0
  the absolute penumbra volume comparison between NBO and control group
volume of core infarction at 4h following randomizing | Day 0
  core infarction volume comparison between NBO and control group
volume of hypoperfusion region hypoperfusion at 4h following randomizing | Day 0
  the volume of hypoperfusion region hypoperfusion comparison between NBO and control group
National Institutes of Health Stroke Scale (NIHSS) score at 24h following randomizing | Day 1
  the comparison of NIHSS score between NBO and control group; NIHSS score ranges from 0 to 42, and higher scores mean a worse outcome.
modified rankin scale (mRS) score at 90 days following randomizing | Month 3
  the mRS score comparison between NBO and control group; mRS score ranges from 0 to 5, and the higher score means a worse outcome.
Barthel Index at 90 days following randomizing | Month 3
  the comparison of Barthel Index between NBO and control group
EQ-5D index at 90 days following randomizing | Month 3
  the comparison of EQ-5D index between NBO and control group
BBB injured biomarkers at baseline and 24h following randomizing | Day 1
  the levels of BBB injured biomarkers comparison between NBO and control group
Cerebral oxygen concentration at baseline and 4h following randomizing | Day 0
  the levels of cerebral oxygen comparison between NBO and control group

CONTACTS AND LOCATIONS:
Overall Officials: Xunming Ji, MD, Principal Investigator — Xuanwu Hospital of Capital Medical University
Locations (1):
- Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China